CLINICAL TRIAL: NCT07341438
Title: Physical Activity in the Management of Personality Disorders: Protocol for a Three-Arm Randomized Feasibility Trial (The PANDA Trial)
Brief Title: Physical Activity in the Management of Personality Disorders
Acronym: PANDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Midtgaard (Other)
Collaborators: Danish Council for Independent Research (Other); Helsefonden, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Julie Midtgaard, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Organization: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-25047904
Record Dates: First submitted 2025-12-12; First posted 2026-01-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Borderline Personality Disorder (BPD); Avoidant Personality Disorders
Keywords: Physical activity; karate; walking; pedometer; martial arts; psychiatry; personality disorders; borderline personality disorder; avoidant personality disorder; feasibility; rct; randomized controlled trial; exercise
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual (Active Comparator): Participants in this arm receive treatment as usual and function as the control group.
  Interventions: Other: Treatment as usual (TAU)
- Karate (Experimental): Participants receive supervised karate training twice a week for 8 weeks from experienced instructors.
  Interventions: Behavioral: Karate; Other: Treatment as usual (TAU)
- Walking (Experimental): Participants follow an 8-week pedometer-based walking program with individually tailored goals.
  Interventions: Behavioral: Pedometer-based walking; Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Karate — The karate group will be offered an 8-week, group-based Shotokan Karate-Do program with two 1-hour sessions per week, delivered at a local karate club. Sessions will be led by two experienced instructors who has recieved lectures in relevant personality pathology and treatment principles. The instructors will plan and adapt the training, which includes meditation to promote focus and calm, Kihon (basic techniques) to practice fundamental movements, Kumite (partnered exercises) to develop coordination, collaboration, and controlled sparring skills, and stretching to support recovery and flexibility. Exercises will be tailored individually to participants' needs, addressing both physical and cognitive aspects of training. Participants will receive relevant equipment, such as a karate uniform and participants may continue attending classes after the 8-week intervention until the end of the study.
  Arms: Karate
Behavioral: Pedometer-based walking — The pedometer-based walking group include a pedometer (Garmin VivoFit 4) and a walking diary, inspired by NICE guidance (PH41). Materials will be reviewed with each participant to ensure understanding and support individual goal-setting. Goals will be tailored to each participant, aiming either to gradually increase daily PA or to establish a structured and manageable activity routine, depending on individual needs and preferences. The diary encourages daily step recording and reflection on physical activity habits. Throughout the 8-week intervention, participants will receive regular check-ins by phone or online at weeks 2, 4, and 6 to review progress, provide structured feedback, and adjust goals as needed.
  Arms: Walking
Other: Treatment as usual (TAU) — Treatment as usual comprise treatment as usual within the psychiatric services. Participants are engaged in ongoing psychotherapeutic treatment when referred to the PANDA study, which includes group and/or individual therapy. As part of the group allocation information, they will be informed about the official Danish physical activity guidelines. Participants will be encouraged to continue their usual daily activities without any specific guidance toward or restriction from engaging in other interventions.

SUMMARY:
The PANDA trial is studying whether two types of physical activity - a walking program and supervised karate training - are safe, acceptable, and possible for adults with certain personality disorders. The goal is to see if these activities can help people while being safe and easy to do.

Who can take part:

* Adults with borderline personality disorder or avoidant/anxious personality disorder.
* People receiving treatment at two outpatient mental health clinics in the Capital Region of Denmark.
* The study plans to include about 60 participants.

What will happen in the study:

Participants are randomly assigned to one of three groups:

* Usual treatment only (control group).
* Usual treatment plus walking program: an 8 - week pedometer - based program with goal setting and follow-up sessions.
* Usual treatment plus supervised karate training: an 8 - week program led by experienced instructors.

What the study will look at:

* Main goal: Check if the programs can be done as planned, including whether participants attend sessions, follow the program, and stay safe.
* Other outcomes: Possible changes in physical health, fitness, emotions, personality symptoms, body image, and daily activity.
* Data will be collected through physical tests, questionnaires, and follow-up interviews about participants' experiences and motivation.
* Measurements will take place at the start, after 8 weeks, and after 12 weeks (follow-up questionnaires only).

Why this study is important:

The results will help researchers decide if it is possible to run a larger study in the future to see if walking or karate training can improve health and wellbeing for people with personality disorders.

DETAILED DESCRIPTION:
OBJECTIVE: The PANDA trial aims to examine the feasibility, acceptability and safety of two physical activity (PA) interventions - pedometer-based walking combined with treatment as usual and karate training combined with treatment as usual - compared to treatment as usual alone. The trial will also explore a range of secondary objective and subjective outcomes. The specific objectives are to:

1. Assess feasibility for a future full-scale trial by measuring screening, recruitment, retention and attendance rates, and intervention safety.
2. Describe changes in objective (body composition and physical fitness) and subjective (patient-reported measures of emotion regulation, personality disorder symptoms and severity, interpersonal functioning, personal recovery, PA behavior, body awareness, and body image) outcomes within and between groups, to estimate the standard deviation of each outcome to inform sample size calculations for a future definitive trial.
3. Explore participant experiences using qualitative methods to assess acceptability and perceived impact of the interventions.

RECRUITMENT: Participants will be recruited from two psychotherapeutic clinics. Eligible patients will be identified during routine treatment by clinical staff based on predefined criteria. Staff will provide brief information about the trial and refer interested individuals to the research team. Additionally, potential participants may self-refer in response to posters in the two clinics. However, all self-referred patients must still meet the trial's inclusion criteria.

Detailed information about the study will then be provided in an information session, which can be conducted either in person or via telephone. Participants will have the option to be accompanied by a support person during this session. A minimum of 24 hours will be provided for reflection before scheduling the baseline visit. At the baseline visit, written informed consent will be obtained prior to any study assessments. Recruitment will continue until 60 participants are included or until July 1, 2026, whichever comes first. If fewer than 20 participants are recruited by April 1, 2026, the study will proceed as a non-randomized trial, allowing participants to select their preferred intervention arm.

STUDY VISITS: Participants will be assessed at three time points: baseline, 8 weeks, and 12 weeks. Baseline and 8-week assessments will be conducted in person, including completion of self-report questionnaires and physical measurements (body composition and cardiorespiratory fitness). The 12-week follow-up consists of questionnaires only and can be completed online at home via REDCap, with no in-person visit required.

After completing the 12-week follow-up (T2), participants originally assigned to the control or walking groups may choose to join the karate program if they wish.

SAMPLE SIZE: The trial aims to include a total of 60 participants, with 20 per arm, adhering to the sample size recommendations for feasibility and pilot trials which suggest that 15 to 25 participants per arm are needed to detect small to medium effect sizes in a subsequent main (definitive) trial with 90% power and 5% significance.

RANDOMIZATION: Eligible participants who provide written informed consent will be randomized 1:1:1 to either treatment as usual (TAU), karate plus TAU (KI+TAU), or pedometer-based walking plus TAU (PI+TAU) after the baseline assessment. Randomization will be performed using a computer-generated list created in the statistical software R and managed in Research Electronic Data Capture (REDCap) by a member of the research team not involved in the PANDA trial, ensuring that allocation remains concealed from PANDA study personnel. Randomization will be conducted in blocks of three and six throughout the study. This approach ensures that the karate intervention can start as a group of six once a total of 18 participants have been randomized, providing six participants in each study arm. Thereafter, inclusion will continue on a rolling, slow-open basis.

ANALYTICAL PLAN:

Analysis will be primarily descriptive. Quantitative outcomes will be summarized using standard methods for rates, proportions, percentages, and sample means, with means, standard deviations, and 95% confidence intervals reported for secondary outcomes at baseline, 8-week, and 12-week follow-ups for each group. Participants will be analyzed according to their allocated group regardless of post-randomization behavior (i.e., intention-to-treat analysis). Missing data will be reported, and no imputation will be performed for feasibility outcomes.

QUALITATIVE SUB-STUDY: Postintervention semi-structured individual interviews will be conducted with participants in the intervention groups. In addition, participants who withdraw from the trial will be invited to take part in an interview. An interview guide, informed by theoretical frameworks on motivation for health behavior change and the theoretical framework of acceptability including affective attitude, burden, perceived effectiveness, ethicality, intervention coherence, opportunity costs, and self-efficacy will be used to explore participants' experiences of the interventions, perceived value, and barriers to engagement. Participants will be purposefully sampled. The investigators estimate that 7-8 interviews per intervention arm will be sufficient. However, the final sample size will be assessed continuously and guided by the concept of information power. Qualitative data from participant interviews will be analyzed using reflexive thematic analysis as described by Braun and Clarke, and all analyses will be conducted using appropriate software.

SAFETY: The trial will be conducted in accordance with the Declaration of Helsinki (2008), and adverse events (AEs) and serious adverse events (SAEs) will be defined according to International Council for Harmonisation - Good Clinical Practice (ICH-GCP). All participants will complete bi-weekly online questionnaires to report AEs related to the interventions, such as minor sports-related injuries during karate sessions or signs of psychological strain. Mild fatigue or lightheadedness may occur during the submaximal cycling test. Bioimpedance assessment is non-invasive, conducted according to manufacturer guidelines, and excludes participants with contraindications (e.g., pregnancy, pacemaker). Karate instructors and research staff are trained to recognize warning signs of distress or escalating tension and to respond according to predefined safety procedures. SAEs will be reported immediately to the principal investigator (JMi) and trial physician (PV), with intervention-related SAEs also reported to the Ethics Committee. Participants are monitored until resolution, with coverage provided by the Danish Patient Compensation Scheme and karate-related injuries covered by the Danish Karate Federation.

PPI: Three advisors with lived experience are involved from the inception of the PANDA trial, contributing to safety considerations, trial procedures, and the refinement and piloting of questionnaires, participant materials, and trial equipment. During the trial, advisors with lived experience will offer general guidance to support the conduct of the study and help ensure that participant perspectives are considered throughout. They will also contribute to the interpretation and communication of study results.

ETHICS: The trial follows the ethical principles of the Declaration of Helsinki and the standards of the ICH-GCP. The protocol has been approved by the Ethics Committee for the Capital Region of Denmark (H-25047904, protocol version 6) and reviewed by the Capital Region of Denmark's Research Legal Office (p-2025-20202). The study complies with the General Data Protection Regulation (GDPR) and the Data Protection Act.

Any changes to the protocol will be documented in protocol amendments, which must be approved by the Ethics Committee for the Capital Region of Denmark and reported when the study is disseminated.

The risk of serious adverse events is expected to be low. Minor adverse effects related to the interventions may occur, and appropriate monitoring will be in place to ensure participant safety. The anticipated benefits of the interventions justify conducting the trial.

FINANCES, INTEREST OF CONFLICTS AND PARTICIPANT COMPENSATION:

The PANDA Trial is funded by the Danish Council for Independent Research (DKK 1,924,524; grant number 4309-00019B) and Helsefonden, Denmark (DKK 200.000; grant number 25-B-0171). The fundings are administered through the Mental Health Centre Glostrup, covering all trial-related costs. The funders had no role in the trial design and will have no role in its conduct, analysis, reporting, or ethical oversight.

The investigators report no conflicts of interest. Participants are compensated in accordance with the guidelines of the Danish National Committee on Health Research Ethics: karate group members receive access to the 8-week program and may keep the uniform, while walking group participants receive a pedometer. Travel expenses for in-person assessments or karate sessions may be reimbursed, with no additional financial incentives offered.

DISSEMINATION: Qualitative, and quantitative results, including feasibility outcomes assessed at weeks 0, 8, and 12, will be reported in separate publications. Affect (Positive and Negative Affect Schedule [PANAS]) will be reported separately in an independent publication, following the publication of the primary and other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years)
* documented diagnosis of borderline personality disorder (BPD; F60.3, ICD-10) or avoidant personality disorder (AVPD; F60.6, ICD-10), as confirmed in the patient's medical record.
* at the time of recruitment, participants must be receiving treatment at one of two specialized psychotherapeutic outpatient clinics (Clinic A or Clinic B) in the Capital Region of Denmark
* proficient in Danish.

Exclusion Criteria:

* Individuals with a documented diagnosis of antisocial personality disorder (F60.2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Referral rate (initial interest rate) | Assessed continuously throughout the recruitment period.
  The proportion of patients approached by clinical staff who agree to be referred to the research team for further information about the study.
  Calculation: Number of patients referred to the research team/Number of patients approached by clinical staff.
Screening rate | Assessed continuously throughout the recruitment period, prior to each participant's baseline assessment.
  The proportion of participants referred by clinical staff who complete the research team's information session.
  Calculation: Number of participants attending the information session/Number of participants referred by clinical staff.
Recruitment rate (consent rate) | Assessed continuously throughout the recruitment period.
  The proportion of participants who consent to join the trial after attending the research team's information session.
  Calculation: Number of participants providing informed consent/Number of participants attending the information session.
Retention rate | From each participant's baseline assessment (week 0) to their 12-week follow-up.
  The proportion of participants who remain in the trial until completion.
  Calculation: Number of participants completing the study/Number of participants initially enrolled.
Adherence | Assessed during the 8-week intervention period for each participant.
  The extent to which participants comply with their assigned intervention.
  Individual criteria:
  Karate group: Attendance at ≥8 of 16 sessions (≥50%). Walking group: Achievement of individually defined weekly step goals in ≥6 of 8 weeks (≈70%).
  Progression criterion: Progression to a full-scale RCT without modification requires that at least 70% of participants in each intervention arm meet these adherence criteria.
Safety (Adverse Events) | Weeks 0-8 for the intervention period for each participant; medical record review extend through 12-week follow-up.
  Occurrence of any adverse events (AEs) during the intervention period.
  Assessment:
  Bi-weekly self-reported electronic questionnaires via REDCap. Extraction from medical records for events such as emergency department visits.
Reasons for non-participation or drop-out | Collected throughout recruitment and study participation for each individual (from invitation to 12-week follow-up).
  Documented explanations provided voluntarily by participants who decline participation or discontinue the trial.
  Assessment: Categorized according to predefined options (e.g., intervention not attractive, inconvenient timing, travel distance, lack of energy, other).

SECONDARY OUTCOMES:
Simple Physical Activity Questionnaire (SIMPAQ) | Baseline and 8-weeks follow-up.
  What it measures: Physical activity behavior and sedentary behavior over the previous 7 days.
  Administration: Clinician-administered structured interview.
  Score range: Continuous estimates in minutes per day for each activity category (sleep, sedentary behavior, walking, structured exercise, other physical activity).
  Direction: Higher values on physical activity measures (e.g., walking or exercise) indicate greater activity, whereas higher values on sedentary behavior measures indicate more inactivity.
Exercise Addiction Inventory (EAI) | Baseline, 8 weeks, and 12 weeks follow-up.
  What it measures: Risk of exercise addiction, including compulsive exercise, loss of control, tolerance, and negative impacts on life.
  Administration: Self-report questionnaire. Participants respond to each of the 6 items by selecting one statement on a 5-point scale:
  1 = Strongly disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Strongly agree
  Scoring: 6 items × 1-5 points each. Total score is obtained by summing all items. Score range: 6-30.
  Direction: Higher scores indicate greater risk of exercise addiction.
Body composition | Baseline and at 8-weeks follow-up.
  Body composition, including fat mass and muscle mass, will be assessed using bioelectrical impedance analysis with the Seca mBCA 515 (Seca, Hamburg, Germany; Approval type: BCA01A, DE-21-nawid-ptb009). Outcomes will be reported both as absolute values in kilograms (kg) and as relative values expressed as a percentage of total body weight. All measurements will be conducted in accordance with standardized procedures and with regular device calibration.
Personality Disorder Severity Scale - ICD 11 (PDS ICD 11) | Baseline, 8 weeks, and 12 weeks follow up.
  What it measures: Severity of personality dysfunction, including impairments in self functioning, interpersonal functioning, emotional regulation, and psychosocial functioning.
  Administration: Self report questionnaire (14 items).
  Scoring:
  Items 1-10 are scored 2 - 1 - 0 - 1 - 2 and items 11-14 are scored 0 - 1 - 2 - 3. The total score is the sum of all 14 items, yielding a range from 0 to 32.
  Direction: Higher scores indicate greater severity of personality dysfunction.
Inventory of Interpersonal Problems - 32 items (IIP 32) | Baseline, 8 weeks, and 12 weeks follow up.
  What it measures: Distress associated with interpersonal difficulties, including problems in assertiveness, sociability, and overly accommodating behaviors.
  Administration: Self report questionnaire.
  Scoring: Respondents rate each of the o 32 items, each rated on a 5-point Likert scale: 0 = Not at all, 1 = A little bit, 2 = Moderately, 3 = Quite a bit, 4 = Extremely. All item scores are summed to form a total score.
  Score range is 0 -128 (32 items × 4).
  Direction: Higher scores indicate greater interpersonal problems or distress.
Questionnaire about the Process of Recovery (QPR) | Baseline, 8 weeks, and 12 weeks follow-up.
  What it measures: Personal recovery, including empowerment, hope, and self-perception.
  Administration: Self-report questionnaire (15 items).
  Scoring:
  Each item is rated on a 5-point scale: 0 = Strongly disagree, 1 = Disagree, 2 = Neither agree nor disagree, 3 = Agree, 4 = Strongly agree.
  Total score is the sum of all 15 items. Score range: 0-60.
  Direction: Higher scores indicate greater personal recovery.
Difficulties in Emotion Regulation Scale - 16 items (DERS 16) | Baseline, 8 weeks, and 12 weeks follow-up.
  What it measures: Difficulties in emotion regulation, including awareness, understanding, acceptance of emotions, and ability to control impulses and use strategies to regulate emotions.
  Administration: Self-report questionnaire. Scoring: 16 items, each rated on a 5-point scale: 1 = Almost never, 2 = Sometimes, 3 = About half the time, 4 = Most of the time, 5 = Almost always Total score is obtained by summing all items. Score range: 16-80.
  Direction: Higher scores indicate greater difficulties in emotion regulation.
Positive and Negative Affect (PANAS) | Baseline, 8 weeks, and 12 weeks follow-up.
  What it measures: Intensity of positive and negative emotions, such as alertness, enthusiasm, nervousness, and distress.
  Administration: Self-report questionnaire.
  Scoring: 20 items (10 positive affect, 10 negative affect), each rated on a five-point scale: 1 = very slightly or not at all, 2 = a little, 3 = moderately, 4 = quite a lot, 5 = extremely.
  Separate total scores are calculated for positive and negative affect. Score range: 10 to 50 for each subscale (10 items × 1-5).
  Direction: Higher positive affect scores indicate greater positive emotions; higher negative affect scores indicate greater negative emotions.
BSL 23 Supplementary Items (from the Borderline Symptom list (BSL-23)) | Baseline, 8 weeks, and 12 weeks follow-up.
  What it measures: Frequency of self-destructive behaviors, including impulsive, high-risk, and self-harming behaviors (Only the supplementary items from the BSL 23 that assess the number of episodes of each behavior are included).
  Administration: Self-report questionnaire.
  Scoring: 6 items, each rated on a five-point scale: 0 = Not at all, 1 = Once, 2 = 2-3 times, 3 = 4-6 times, 4 = Daily or more often.
  Total score is obtained by summing all items. Score range: 0 to 24 (6 items × 4).
  Direction: Higher scores indicate greater frequency of self-destructive behaviors.
The Body Appreciation Scale 2 (BAS-2) | Baseline, 8 weeks, and 12 weeks follow-up.
  What it measures: Positive body image, including acceptance, respect, and appreciation of one's body.
  Administration: Self-report questionnaire. Participants are asked to indicate how often each statement is true for them.
  Scoring: 10 items, each rated on a five-point Likert scale: 1 = Never, 2 = Seldom, 3 = Sometimes, 4 = Often, 5 = Always.
  Total score is obtained by summing all items. Score range: 10 to 50 (10 items × 5).
  Direction: Higher scores indicate greater body appreciation.
The Multidimensional Assessment of Interoceptive Awareness (MAIA) - Self-Regulation subscale | Baseline, 8 weeks, and 12 weeks follow-up.
  What it measures: Ability to regulate stress or emotional distress through attention to bodily sensations (interoceptive self-regulation).
  Administration: Self-report questionnaire. Participants indicate how often each statement is true for them.
  Scoring: Self-Regulation subscale consists of 4 items (S23, S24, S25, S26), each rated on a 6-point numeric scale: 0 = Never, 1, 2, 3, 4, 5 = Always.
  Total score is obtained by averaging the 4 items. Score range: 0 to 5 (average of 4 items).
  Direction: Higher scores indicate greater ability to regulate stress or emotional distress via body awareness.
Body Awareness Scale - Experience (BAS-E) (from the Body Awareness Scale - Movement Quality and Experience (BAS MQ E)) | Baseline, 8 weeks, and 12 weeks follow-up.
  What it measures: Subjective bodily awareness and experiences, including posture, movement, muscle tension, pain, breathing, appearance, functional limitations, and engagement in movement over the past week.
  Administration: Self-report questionnaire.
  Scoring: Item 1: Free-text response describing bodily sensations in participant's own words.
  Items 2-7: participants select one of four statements per item, ranging from more positive to more negative experiences.
  Item 8: Yes/No response. Item 9: Multiple-choice; participants can select all statements that apply.
  Directions: Items 2-7, higher scores indicate more negative experiences or greater functional limitations. Items 1, 8, and 9 are used descriptively.
Cardiorespiratory fitness (VO₂max) | Baseline and at 8-weeks follow-up
  Aerobic and cardiorespiratory fitness will be estimated using the submaximal revised Ekblom-Bak cycle ergometer test performed on a Monark Ergomedic 828 E (Monark, Sweden). The test provides an estimate of maximal oxygen uptake (VO₂max, mL·kg-¹·min-¹) based on heart rate response to standardized submaximal workloads. The ergometer will be calibrated and individually adjusted according to standardized procedures. Higher estimated VO₂max values indicate greater aerobic and cardiorespiratory fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Midtgaard, Professor, Principal Investigator — Copenhagen University Hospital - Amager and Hvidovre
Locations (2):
- Denmark (2):
  - Mental Health Center Stolpegård, Copenhagen University Hospital -Mental Health Services CPH, Copenhagen Denmark, Gentofte Municipality, Capital Region
  - Mental Health Centre Glostrup, Copenhagen University Hospital - Amager and Hvidovre, Denmark, Glostrup Municipality, Capital Region

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared publicly due to ethical constraints; however, qualified researchers may submit individual requests for access.

REFERENCES:
- [Background] Petersen J, Palic S, Nyboe L, Schuster M, Videbech P, Midtgaard J. Physical activity in the management of borderline personality disorder: A scoping review. Psychiatry Res. 2025 Aug;350:116535. doi: 10.1016/j.psychres.2025.116535. Epub 2025 May 5. PMID 40398190